CLINICAL TRIAL: NCT01731340
Title: The Effect of Dietary Calcium Intake as Compared to Calcium Supplementation on Vascular Health and Bone Health in Postmenopausal Women
Brief Title: A Study on the Impact of Calcium on Woman's Vascular Health
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Suzanne Morin, MD MSc FRCP, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GEN-11-231
Record Dates: First submitted 2012-11-16; First posted 2012-11-21 (Estimated); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Cardiovascular Diseases; Osteoporosis
Keywords: Calcium Supplements; Dairy Foods; Cardiovascular Diseases; Osteoporosis; Postmenopause; Vitamin D; Micronutrients; Primary Prevention; Bone Health
MeSH Terms: conditions — Cardiovascular Diseases; Osteoporosis | interventions — Calcium Citrate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Supplemental Calcium (Active Comparator): * 750 mg Calcium Citrate per day
  * 800 IU Vitamin D3 per day
  * Low Dietary Calcium (450 mg per day)
  Interventions: Dietary Supplement: Calcium Citrate; Other: Low Dietary Calcium
- Dietary Calcium (Active Comparator): * 400 IU Vitamin D3 per day
  * High Dietary Calcium (1200 mg per day)
  Interventions: Other: High Dietary Calcium
- Usual Diet (No Intervention): * 400 IU Vitamin D3 per day
  * Unrestricted Dietary Calcium

INTERVENTIONS:
Dietary Supplement: Calcium Citrate — 750mg
  Arms: Supplemental Calcium
Other: Low Dietary Calcium — 450 mg
  Arms: Supplemental Calcium
Other: High Dietary Calcium — 1200 mg
  Arms: Dietary Calcium

SUMMARY:
The overarching aim of this randomized clinical trial is to estimate the effect of dietary intake of calcium as compared to supplemental calcium on the vascular system and markers of vascular and bone health in postmenopausal women.

DETAILED DESCRIPTION:
Calcium and vitamin D are essential nutrients for optimal bone health throughout life. Research has shown that postmenopausal women who consume appropriate amounts of these nutrients have better bone strength and fewer fractures than those who don't. However, researchers have recently questioned the safety of calcium and vitamin D obtained through supplements as they might increase the risk of cardiovascular events such as heart attacks and strokes.

The investigators propose to estimate the effect of dietary intake of calcium as compared to supplemental calcium on vascular and bone health in postmenopausal women.

Eligible participants will be assigned by chance (like a coin toss) to one of three groups: (1) 1200 mg of calcium from dietary sources and 1 capsule of 400 IU vitamin D supplement everyday after the first meal of the day; (2) 450 mg of calcium from dietary sources, 2 tablets of 250 mg calcium citrate supplement and 1 capsule of 800 IU vitamin D supplement everyday after the first meal of the day and 1 tablet of 250 mg calcium citrate supplement after the evening meal or snack; or (3) unrestricted calcium from dietary sources and 1 capsule of 400 IU vitamin D supplement everyday after the first meal of the day. Participants have an equal chance of being assigned to any of these three groups until 26 participants have been assigned to group (3). At this time participants will continue to be assigned by chance to either of the two remaining groups only.

Participants will also attend appointments at the Montreal General Hospital every 6-months where they will undergo anthropometric measurements, blood tests, urine tests, non-invasive ultrasounds to measure arterial stiffness and questionnaires. The questionnaires ask about health; lifestyle habits such as physical exercise, diet, and smoking; use of medications and dietary supplements; family history of illness, and past medical diagnoses. Participants will also receive monthly phone calls from study staff to monitor for adverse events and adherence.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 50 or more
* 2 years since last menstrual period
* Body Mass Index between 20 and 35 kg/m2

Exclusion Criteria:

* Atrial Fibrillation
* Coronary artery disease
* Myocardial infarction
* Stroke
* Transient ischaemic attack
* Peripheral vascular disease
* Sleep apnea
* Hypertension
* Hyperlipidemia
* Hyperparathyroidism
* Urinary tract lithiasis
* Rheumatoid arthritis
* Crohn's disease
* Ulcerative colitis
* Short gut syndrome
* Celiac disease
* Diabetes
* Cancer (any other than basal cell cancer of the skin)
* Pre-eclampsia
* Smoked in the last 5 years
* Cocaine use in the last year
* Consumption of more than 9 alcoholic drinks per week
* Chronic NSAID use
* Use of oral glucocorticoids or HRT (excluding vaginal preparations) in the last 2 years
* Use of anti-osteoporosis medications (bisphosphonates, selective estrogen-receptor modulators, denosumab, teriparatide, or calcitonin) in the last 3 years or anti-osteoporosis therapy which ended more than 3 years ago and whose duration was ≥ 5 years, or a fracture of the spine, shoulder, or hip was sustained while therapy
* Use of calcium and vitamin D supplements (including multivitamins and calcium-containing antacids) in the last 2 months
* High 10-year probability of major osteoporotic fracture (FRAX without BMD > 20%)

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2018-11-14 (Actual); Study Completion 2018-11-14 (Actual)

PRIMARY OUTCOMES:
Vascular System | 12 months
  Measured as changes in:
  * Arterial stiffness (carotid-femoral pulse wave velocity)
  * Arterial wall thickness (carotid intima-media thickness)

SECONDARY OUTCOMES:
Hemodynamics | 12 Months
  Measured as changes in:
  - Peripheral blood pressure

OTHER OUTCOMES:
Blood Biomarkers | 12 months
  Measured as changes in:
  * Vascular health biomarkers
  * Bone health biomarkers
Anthropomorphic measurements | 12 months
  Measured as changes in bone health biomarkers.
  * Body mass index
  * Waist circumference
  * Body fat %
Adverse Events | 12 months
  Occurrence of cardiovascular, cerebrovascular and renal events as well as fractures and intolerance to interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Morin, MD MSc, Principal Investigator — McGill University Hospital Center
Locations (1):
- Department of Internal Medicine; Montreal General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No